CLINICAL TRIAL: NCT00193973
Title: A Phase 2 Study of Idarubicin Based Combined Modality Therapy in Primary Central Nervous System Lymphoma
Brief Title: Idarubicin Based Combined Modality Therapy in Primary CNS Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Trans Tasman Radiation Oncology Group (Other)
Collaborators: Australasian Leukaemia and Lymphoma Group (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TROG 01.02; ALLG LY4 (Other: ALLG)
Record Dates: First submitted 2005-09-13; First posted 2005-09-19 (Estimated); Last update posted 2017-02-17 (Actual); Status verified 2017-02

CONDITIONS: Primary Central Nervous System Lymphoma
Keywords: Lymphoma; PCNSL; Primary CNS lymphoma
MeSH Terms: conditions — Lymphoma | interventions — Idarubicin; Methotrexate; Filgrastim; Radiotherapy; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Active Comparator)
  Interventions: Drug: Idarubicin, Methotrexate, Filgrastim, intrathecal Ara-C; Radiation: Radiation Therapy

INTERVENTIONS:
Drug: Idarubicin, Methotrexate, Filgrastim, intrathecal Ara-C — Idarubicin 15mg/m2 days 1, 22. Filgrastim 5mcg/kg until neutrophil recovery days 2, 23. Methotrexate 1g/m2 days 15, 36 and 50.
Radiation: Radiation Therapy — Whole brain Irradiation, 30Gy in 20 fractions over 4 weeks
  Other Names: Radiation, Radiotherapy

SUMMARY:
Idarubicin combined with high dose methotrexate and moderate dose radiotherapy will achieve similar survival outcomes but with reduced neurotoxicity compared to regimens using methotrexate with high dose radiotherapy.

DETAILED DESCRIPTION:
Combined modality therapy in PCNSL has improved survival outcomes but at the cost of unacceptable rates of neurotoxicity when high dose radiotherapy is used. Idarubicin has activity in systemic lymphomas and crosses the blood brain barrier and may add to the efficacy of methotrexate. By combining these 2 drugs with moderate dose radiotherapy survival outcomes should be optimal but with lower rates of neurotoxicity.

Comparison: TROG has previously performed a phase 2 study using methotrexate with high dose radiotherapy and this will allow comparison of survival and neurotoxicity rates.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven primary CNS lymphoma.
* Absence of disease outside the CNS.
* ECOG performance status 0-3
* Negative HIV status.
* Peripheral blood counts with granulocytes >1.5 x 109L and platelets > 100 x 109L. Serum creatinine <150mmol/L. Serum bilirubin <1.5 times and AST <2 times upper limit of normal.
* Age >18 and <=70 years.
* Patients must give written informed consent.
* Corticosteroids prior to histological diagnosis are allowed.

Exclusion Criteria:

* Previous history of malignancy (other than non-melanomatous skin carcinoma, or carcinoma in situ of cervix completely excised).
* Patients who are pregnant or lactating.
* NYHA (New York State Heart Association classification) cardiac failure grade 3
* Macroscopic spinal thecal or spinal cord disease.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2001-07; Primary Completion 2008-07 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
To estimate the median and 2 year overall survival. | Estimate of survival at 2 years and at 5 years.

SECONDARY OUTCOMES:
Assess acute toxicity. | Interim actute toxicity analyses will be performed at accrual points: 5, 10, 15, 20 and 25 patients.
Assess functional indices of living in patients with PCNSL. | Analysis will be at 5 years.
To estimate the risk of late neurotoxicity relative to results achieved in TROG 92.01. | Analysis at 3 years.

CONTACTS AND LOCATIONS:
Overall Officials: Peter O'Brien, FRANZCR, Study Chair — Newcastle Mater Misericordiae Hospital
Locations (15):
- Australia (13):
  - The Canberra Hospital, Garran, Australian Capital Territory
  - Calvary Mater Newcastle, Newcastle, New South Wales
  - Prince of Wales Hospital, Randwick, New South Wales
  - Westmead Hospital, Wentworthville, New South Wales
  - Illawarra Cancer Care Centre, Wollongong, New South Wales
  - Royal Brisbane Hospital, Herston, Queensland
  - Mater QRI, South Brisbane, Queensland
  - Premion - Tugun, Tugun, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Andrew Love Cancer Centre, Geelong Hospital, Geelong, Victoria
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
  - Sir Charles Gairdner Hospital, Nedlands, Western Australia
- New Zealand (2):
  - Auckland Hospital, Auckland
  - Christchurch Hospital, Christchurch

REFERENCES:
- See also: Click here for more information about this study on the TROG official website — http://www.trog.com.au